CLINICAL TRIAL: NCT02887820
Title: A Pilot Study in Feasibility and Safety: Point of Care Testing With Thromboelastography (TEG) for Blood Product Transfusion in Patient's Requiring Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Evaluating the Use of Thromboelastography (TEG) in Patient's Requiring Extracorporeal Membrane Oxygenation (ECMO)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A new standard of care was introduced making it impossible to continue with the study. Additionally, some of the blood product and transfusion related outcomes were not collected because this data was not present in the EMR.
Sponsor: Stephen Esper (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Stephen Esper, Assistant Professor of Anesthesiology, Chief of Perioperative Services, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19070239
Record Dates: First submitted 2016-08-25; First posted 2016-09-02 (Estimated); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Heart Disease; Lung Disease
Keywords: ECMO; TEG
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pilot Arm (Other): All subjects enrolled in the trial will be in the pilot group. These subjects will have traditional laboratory coagulation and blood transfusion tests (baseline arterial blood gas (ABG), complete blood count (CBC), fibrinogen, platelet count, aPTT, PT, anti-Xa, ACT), as well as thromboelastograph (TEG). Pertinent TEG results will include: heparinase-kaolin TEG maximum amplitude (MA) in millimeters (mm), heparinase-kaolin TEG r-time in seconds, heparinase-kaolin TEG alpha angle in degrees, and TEG functional fibrinogen (FLEV) MA in mm.
  Interventions: Device: Thromboelastograph

INTERVENTIONS:
Device: Thromboelastograph — A thromboelastograph flowchart will be followed in addition to traditional laboratory tests to manage blood transfusion and coagulation decisions
  Other Names: TEG 5000

SUMMARY:
This is a pilot study that seeks to evaluate the feasibility and safety of using a TEG algorithm in addition to traditional laboratory tests to guide transfusion and coagulation management of ECMO patients.

DETAILED DESCRIPTION:
All adult patients requiring ECMO will be considered for the trial, with a target enrollment of 50 participants over a two-year period. For each enrolled participant, a TEG transfusion algorithm will be followed for patients exhibiting inadequate hemostasis in the operating room (Flowchart 1). Once patient has a normal TEG result with adequate hemostasis, either heparin or bivalirudin will be used as the anticoagulant. If patients are receiving no anticoagulation or heparin anticoagulation then a second TEG algorithm will be followed in the ICU when hemostasis is normal and heparin is introduced (Flowchart 2). If patients are receiving bivalirudin as their anticoagulation strategy, the transfusion parameters with TEG application will not apply. In addition to determining the compliance and feasibility of following these TEG algorithms, clinical outcome data including transfusion rates, types of blood products transfused, estimated blood loss and thrombotic events will be collected for every enrolled patient until they are discontinued from ECMO. Statistical analysis of the primary, secondary and tertiary endpoints of this study will determine the likelihood of exploring future clinical trials involving TEG-driven coagulation and transfusion management of the ECMO population.

ELIGIBILITY:
Inclusion Criteria:

* Patient's requiring ECMO placement

Exclusion Criteria:

* Other than children less than 18 years of age, no one will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Esper, MD, MBA, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oliver WC. Anticoagulation and coagulation management for ECMO. Semin Cardiothorac Vasc Anesth. 2009 Sep;13(3):154-75. doi: 10.1177/1089253209347384. PMID 19767408
- [Result] Esmon CT. The impact of the inflammatory response on coagulation. Thromb Res. 2004;114(5-6):321-7. doi: 10.1016/j.thromres.2004.06.028. PMID 15507261
- [Result] Muntean W. Coagulation and anticoagulation in extracorporeal membrane oxygenation. Artif Organs. 1999 Nov;23(11):979-83. doi: 10.1046/j.1525-1594.1999.06451.x. PMID 10564301
- [Result] Colby CE, Sheehan A, Benitz W, Van Meurs K, Halamek LP, Moss RL. Maintaining adequate anticoagulation on extracorporeal membrane oxygenation therapy: Hemochron Junior Low Range versus Hemochron 400. J Extra Corpor Technol. 2003 Mar;35(1):35-8. PMID 12680494
- [Result] Reiner JS, Coyne KS, Lundergan CF, Ross AM. Bedside monitoring of heparin therapy: comparison of activated clotting time to activated partial thromboplastin time. Cathet Cardiovasc Diagn. 1994 May;32(1):49-52. doi: 10.1002/ccd.1810320112. PMID 8039220
- [Result] Despotis GJ, Summerfield AL, Joist JH, Goodnough LT, Santoro SA, Spitznagel E, Cox JL, Lappas DG. Comparison of activated coagulation time and whole blood heparin measurements with laboratory plasma anti-Xa heparin concentration in patients having cardiac operations. J Thorac Cardiovasc Surg. 1994 Dec;108(6):1076-82. PMID 7983877
- [Result] Afshari A, Wikkelso A, Brok J, Moller AM, Wetterslev J. Thrombelastography (TEG) or thromboelastometry (ROTEM) to monitor haemotherapy versus usual care in patients with massive transfusion. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD007871. doi: 10.1002/14651858.CD007871.pub2. PMID 21412912
- [Result] Shore-Lesserson L, Manspeizer HE, DePerio M, Francis S, Vela-Cantos F, Ergin MA. Thromboelastography-guided transfusion algorithm reduces transfusions in complex cardiac surgery. Anesth Analg. 1999 Feb;88(2):312-9. doi: 10.1097/00000539-199902000-00016. PMID 9972747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Arm
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 47.2 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Blood Management Care Follows a TEG Algorithm 90% of the Time
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 4

2. Secondary Outcome: Number of Transfusions Required While on ECMO
Description: Number of patients who required transfusions
Time Frame: From the time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 9

3. Secondary Outcome: Number of Participants That Experience Bleeding or Thrombotic-related Adverse Events, Including Deep Venous Thrombosis or Pulmonary Embolus
Description: Number of patients who experienced bleeding while on ECMO
Time Frame: From the time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 11

4. Secondary Outcome: Chest Tube Output and Overall Estimated Blood Loss
Description: Average chest tube output
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Mean (Full Range); unit: ML
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
ML | 2692 [0 to 8980]

5. Secondary Outcome: Time Between Transfusions
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Population: Data not collected-- the transfusion times are not well documented in the EMR. It is impossible to tell what time transfusions occurred. This data was not collected and the study status was changed to "terminated"
Arm/Group | Pilot Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Type of Blood Products Transfused
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Population: Type of blood products administered is not well documented in the EMR. This data was not collected and the study status was changed to "terminated". DATA NOT COLLECTED, this information does not exist in the EMR. We did not anticipate this at the beginning of the study.
Arm/Group | Pilot Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Pump Exchanges Required
Description: Number of participants who required pump exchanges
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 4

8. Secondary Outcome: Oxygenator Exchanges
Description: NUmber of participants who required oxygenator exchanges while on ECMO
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Population: Data not analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 3

9. Secondary Outcome: Occurrence of Pump Circuit Clotting and Clots in the Oxygenator (Visible Clot Which Did Not Require Circuit/Pump Exchange)
Description: Number of participants with pump circuit clotting
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 2

10. Secondary Outcome: Time to Weaning From/Removal of ECMO
Description: Average time to ECMO removal
Time Frame: From time patient is placed on ECMO until time to weaning from ECMO
Measure: Mean (Full Range); unit: minutes
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
minutes | 19315 [2104 to 54090]

11. Secondary Outcome: Need for Surgical Intervention for Hemorrhage
Description: Number of participants
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm
Number analyzed (Participants) | 15
Participants | 9

12. Secondary Outcome: Specimen Turn Around Time for Lab Tests (CBC, ACT, PT, PTT, Anti-Xa, INR, Platelet Count) and TEG Results
Time Frame: From time patient is placed on ECMO to 30-days post ECMO initiation
Population: This data is not well documented in the EMR. This data was not collected and the study status was changed to "terminated". DATA NOT COLLECTED. NO resources to data mine this information.
Arm/Group | Pilot Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For the duration of time the participant is on ECMO (24 hours to 6 weeks)
Arm/Group | Pilot Arm
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02887820/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02887820/ICF_001.pdf